CLINICAL TRIAL: NCT03148847
Title: Evaluation of Professional Practices on the Management of Cardiogenic Pulmonary Edema (RENAU-OAP)
Brief Title: Management of Cardiogenic Pulmonary Edema (RENAU-OAP)
Acronym: RENAU-OAP
Status: Terminated | Type: Observational
Why Stopped: Only the first part of the study was done.
Sponsor: Centre Hospitalier Annecy Genevois (Other)
Responsible Party: Sponsor
Other Study IDs: 2014-RENAU-1
Record Dates: First submitted 2017-05-02; First posted 2017-05-11 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Dyspnea, Paroxysmal; Heart Failure, Left Sided
MeSH Terms: conditions — Dyspnea, Paroxysmal; Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Baseline care: Patients treated for Cardiogenic Pulmonary Edema into the Northern French Alps Emergency Network between January 1, 2013 and December 31, 2013
  Interventions: Other: Baseline care
- Referential's dissemination: Patients treated for Cardiogenic Pulmonary Edema into the Northern French Alps Emergency Network between January 1, 2017 and December 31, 2017, after referential's dissemination for management of patients with paroxysmal dyspnea due to left sided heart failure
  Interventions: Other: Referential's dissemination

INTERVENTIONS:
Other: Baseline care
  Groups: Baseline care
Other: Referential's dissemination
  Groups: Referential's dissemination

SUMMARY:
The prevalence of heart failure is estimated to 2.3 percent of the adult population and strongly increases with age, according to french disability-health surveys. In France, more than 32,000 annual deaths are attributable to heart failure and the five-year survival rate is similar to those found in many cancers. A better therapeutic management (angiotensin converting enzyme inhibitor and beta-blockers) helped reduce mortality after an episode of heart failure requiring hospitalization, but, nevertheless it remains high.

The severity of cardiogenic pulmonary edema depends on several factors such as etiology, hemodynamic status, effect on hematosis, and fatigue.

It is important to note that cardiogenic pulmonary edema initial management is decisive. In addition, early and adapted management of cardiogenic pulmonary edema is associated with a shorter hospital stay and reduced hospital mortality.

The Coronary Emergency Network (RESURCOR) within the Northern French Alps Emergency Network (RENAU) is an emergency care system structured in the departments of Isère, Savoie and Haute Savoie. Its main goal is to help improve emergency management by using regional good practice guidelines (www.renau.org). In this context, projects aiming to evaluate professional practices are developed regularly. Since emergency management of cardiogenic pulmonary edema has not been evaluated, the Northern French Alps Emergency Network offers an approach to improve professional practices by defining and disseminating guidelines on cardiogenic pulmonary edema management which will then be assessed.

DETAILED DESCRIPTION:
The prevalence of heart failure is estimated to 2.3 percent of the adult population and strongly increases with age, according to disability-health surveys in France. In recent years, effective treatments (revascularization in percutaneous coronary intervention, circulatory assistance) helped reduce mortality in post-myocardial infarction, which combined with the increase of life expectancy has led to an increase number of patients with chronic heart failure. More than 32,000 annual deaths are attributable to heart failure and the five-year survival rate is similar to those found in cancers of the breast, bladder, colon, ovarian, and prostate. A better therapeutic management (angiotensin converting enzyme inhibitor and beta-blockers) helped reduce mortality after an episode of heart failure requiring hospitalization, but, nevertheless it remains high.

Main clinical manifestations are those of left heart failure, such as cardiogenic pulmonary edema which is a medical emergency. Treatment must take into account pathophysiological aspects of heart failure, etiologies of cardiogenic pulmonary edema and any potential factors or triggers apart from general measures. Two consensus statements and an international recommendation help define therapeutic strategies in this particular situation.

Signs suggestive of cardiogenic pulmonary edema include orthopnea, bilateral crackles or wheezing (patients over 70 years without known asthma), edema of the lower limbs, and gallop sound on heart auscultation. The evolution of these signs makes it particularly possible to manage the response to the treatment. The severity of cardiogenic pulmonary edema depends on several factors such as etiology (ECG analysis and chest pain assessment for acute coronary syndrome), hemodynamic status (blood pressure, heart rate), effect on hematosis (cyanosis, oxygen saturation), and fatigue (low respiratory rate with persistent cardiogenic pulmonary edema signs). The respiratory rate represents a simple clinical feature that can be used to quantify dyspnea (sign of severity if greater than 30 per minute in adults) and then follow its evolution (improvement, exhaustion). Disorders of consciousness can testify to the severity of the hemodynamic state and/or exhaustion.

Cardiogenic pulmonary edema management without shock implies urgent administration of vasodilators (trinitrin) and intravenous loop diuretics in presence of congestion signs along with the establishment of a system of care adapted to severity (Emergency Mobile Services or ambulance, hospitalization in Intensive Care Unit, intensive cardiology unit, cardiology or medicine department, or emergency passage). The subsequent therapeutic management will especially depend on initial treatment by the primary care physician, so it is preferable to record doses and hours of medications. Non-hospitalization must remain exceptional for non-severe decompensation with rapidly favorable evolution.

The French Observatory of Acute Heart Failure (OFICA) including nearly 1,800 patients specified epidemiological and therapeutic data of patients hospitalized for cardiogenic pulmonary edema in 2009. However, this study did not describe the initial management of the Mobile Emergency and Resuscitation Service and emergency services of hospitals. It is important to note that cardiogenic pulmonary edema initial management is decisive. In addition, early and adapted management of cardiogenic pulmonary edema is associated with a shorter hospital stay and reduced hospital mortality.

The Coronary Emergency Network (RESURCOR) within the Northern French Alps Emergency Network (RENAU) is an emergency care system structured in the departments of Isère, Savoie and Haute-Savoie. Its main goal is to help improve emergency management by using regional good practice guidelines (www.renau.org). In this context, projects aiming to evaluate professional practices are developed regularly. Since emergency management of cardiogenic pulmonary edema has not been evaluated, the Northern French Alps Emergency Network offers an approach to improve professional practices by defining and disseminating a guideline on cardiogenic pulmonary edema management which will then be assessed.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* hospitalization during one of the two designed period (either year 2013, or year 2017) in a center belonging to Northern French Alps Emergency Network
* diagnosis of cardiogenic pulmonary edema, or heart failure (either left-sided, congestive or unspecified)

Exclusion Criteria:

* people who refuse to have their health information used will not be included
* people whose care will have begun in a center not belonging to the Northern French Alps Emergency Network

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: As the goal of this study is to analyze common practices, data from the french medicalized information system program will be used to select a study population as exhaustive as possible.
  This program is dedicated to systematic collection of data from hospital stays. Each hospital stay is identified by a unique number and a diagnosis is attributed for each, at the end of every hospital stay. Diagnosis are based on the International Classification of Diseases (ICD-10). At hospital levels, a unique stay number can be related to names and addresses of involved patients.
  French medicalized information system program data are analyzed at a regional and then a national level.
  For this study, cases will be screened if they had a I500, I501 and I509 ICD-10 diagnosis (main or associated).
Sampling Method: Non-Probability Sample
Enrollment: 859 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Change of quality of initial care of patients with cardiogenic pulmonary edema after dissemination of good practice standards | an average of 1 week (length of hospitalization for cardiogenic pulmonary edema)
  Two kinds of predefined quality indicators will be evaluated at different stages of care and compared among the two periods, before and after dissemination of good practice standards, looking for informations in medical charts during the management of patients either care by Mobile Emergency and Resuscitation Services or at emergency departments and in mails at time of hospital discharge).

SECONDARY OUTCOMES:
Patients' description at the onset of cardiogenic pulmonary edema (clinical) | an average of 1 week (length of hospitalization for cardiogenic pulmonary edema)
  Clinical characteristics of patients with cardiogenic pulmonary edema included in the two parts of this observational study (whole population).
Patients' description at the onset of cardiogenic pulmonary edema (biological) | an average of 1 week (length of hospitalization for cardiogenic pulmonary edema)
  Biological characteristics of patients with cardiogenic pulmonary edema included in the two parts of this observational study (whole population).
Patients' description at the onset of cardiogenic pulmonary edema (radiological) | an average of 1 week (length of hospitalization for cardiogenic pulmonary edema)
  Radiological characteristics of patients with cardiogenic pulmonary edema included in the two parts of this observational study (whole population).
Patients' description at the onset of cardiogenic pulmonary edema (echocardiographic) | an average of 1 week (length of hospitalization for cardiogenic pulmonary edema)
  Echocardiographic characteristics of patients with cardiogenic pulmonary edema included in the two parts of this observational study (whole population).
Mortality of patients hospitalized for cardiogenic pulmonary edema | an average of 1 week (length of hospitalization for cardiogenic pulmonary edema)
  number of patients dying during hospitalization for cardiogenic pulmonary edema
Needs for Hospitalization in intensive care units | an average of 1 week (length of hospitalization for cardiogenic pulmonary edema)
  number (and rate) of patients with cardiogenic pulmonary edema, requiring hospitalization in intensive care unit
Needs for respiratory assistance | an average of 1 week (length of hospitalization for cardiogenic pulmonary edema)
  number of patients and kind of respiratory assistance for patients with cardiogenic pulmonary edema
Inter-services transfers | an average of 1 week (length of hospitalization for cardiogenic pulmonary edema)
  number of patients who require transfers from an emergency room (or a cardiology ward) to intensive care units and vice-versa
Length of stay in hospital | an average of 1 week (length of hospitalization for cardiogenic pulmonary edema)
  number of days between arrival and discharge
Re-hospitalizations during the first six months | up to six months
  number of re-hospitalizations during the first six months after the onset of cardiogenic pulmonary edema

CONTACTS AND LOCATIONS:
Overall Officials: Loic BELLE, MD, Study Chair — Centre Hospitalier Annecy Genevois
Locations (1):
- CH Annecy Genevois, Pringy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stewart S, MacIntyre K, Hole DJ, Capewell S, McMurray JJ. More 'malignant' than cancer? Five-year survival following a first admission for heart failure. Eur J Heart Fail. 2001 Jun;3(3):315-22. doi: 10.1016/s1388-9842(00)00141-0. PMID 11378002
- [Background] Mebazaa A, Gheorghiade M, Pina IL, Harjola VP, Hollenberg SM, Follath F, Rhodes A, Plaisance P, Roland E, Nieminen M, Komajda M, Parkhomenko A, Masip J, Zannad F, Filippatos G. Practical recommendations for prehospital and early in-hospital management of patients presenting with acute heart failure syndromes. Crit Care Med. 2008 Jan;36(1 Suppl):S129-39. doi: 10.1097/01.CCM.0000296274.51933.4C. PMID 18158472
- [Background] Heart Failure Society Of America. HFSA 2006 Comprehensive Heart Failure Practice Guideline. J Card Fail. 2006 Feb;12(1):e1-2. doi: 10.1016/j.cardfail.2005.11.005. PMID 16500560
- [Background] McMurray JJ, Adamopoulos S, Anker SD, Auricchio A, Bohm M, Dickstein K, Falk V, Filippatos G, Fonseca C, Gomez-Sanchez MA, Jaarsma T, Kober L, Lip GY, Maggioni AP, Parkhomenko A, Pieske BM, Popescu BA, Ronnevik PK, Rutten FH, Schwitter J, Seferovic P, Stepinska J, Trindade PT, Voors AA, Zannad F, Zeiher A; ESC Committee for Practice Guidelines. ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure 2012: The Task Force for the Diagnosis and Treatment of Acute and Chronic Heart Failure 2012 of the European Society of Cardiology. Developed in collaboration with the Heart Failure Association (HFA) of the ESC. Eur Heart J. 2012 Jul;33(14):1787-847. doi: 10.1093/eurheartj/ehs104. Epub 2012 May 19. No abstract available. PMID 22611136
- [Background] Emerman CL. Treatment of the acute decompensation of heart failure: efficacy and pharmacoeconomics of early initiation of therapy in the emergency department. Rev Cardiovasc Med. 2003;4 Suppl 7:S13-20. PMID 14668696
- [Background] Peacock WF 4th, Emerman CL. Emergency department management of patients with acute decompensated heart failure. Heart Fail Rev. 2004 Jul;9(3):187-93. doi: 10.1007/s10741-005-6128-5. PMID 15809816
- [Background] Rivers E, Nguyen B, Havstad S, Ressler J, Muzzin A, Knoblich B, Peterson E, Tomlanovich M; Early Goal-Directed Therapy Collaborative Group. Early goal-directed therapy in the treatment of severe sepsis and septic shock. N Engl J Med. 2001 Nov 8;345(19):1368-77. doi: 10.1056/NEJMoa010307. PMID 11794169
- [Background] Belle L, Fourny M, Reynaud T, Hammer L, Vanzetto G, Labarere J; RENAU-RESURCOR study investigators. Efficacy and safety of glycoprotein IIb/IIIa receptor antagonists for patients undergoing percutaneous coronary intervention within twelve hours of fibrinolysis. Catheter Cardiovasc Interv. 2011 Sep 1;78(3):376-84. doi: 10.1002/ccd.22825. Epub 2011 Mar 16. PMID 21413113
- [Background] Chacornac M, Baronne-Rochette G, Schmidt MH, Savary D, Habold D, Bouvaist H, Marliere S, Belle L, Machecourt J, Vanzetto G; REseau des URgences CORonariennes (RESURCOR). Characteristics and management of acute ST-segment elevation myocardial infarctions occurring in ski resorts in the French Alps: Impact of an acute coronary care network. Arch Cardiovasc Dis. 2010 Aug-Sep;103(8-9):460-8. doi: 10.1016/j.acvd.2010.09.002. Epub 2010 Oct 30. PMID 21074125
- [Background] Debaty G, Belle L, Labarere J, Fourny M, Torres JP, Savary D, Usseglio P, Menthonnex E, Guenot O, Vanzetto G. [Evolution of strategies of revascularisation in acute coronary syndromes with ST elevation. Analysis of the data of RESURCOR]. Arch Mal Coeur Vaiss. 2007 Feb;100(2):105-11. French. PMID 17474495
- [Background] Ferrier C, Belle L, Labarere J, Fourny M, Vanzetto G, Guenot O, Debaty G, Savary D, Machecourt J, Francois P. [Comparison of mortality according to the revascularisation strategies and the symptom-to-management delay in ST-segment elevation myocardial infarction]. Arch Mal Coeur Vaiss. 2007 Jan;100(1):13-9. French. PMID 17405549
- [Background] Fourny M, Belle L, Labarere J, Senee D, Savary D, Debaty G, Vanzetto G, Francois P. [Analysis of the accuracy of a coronary syndrome register]. Arch Mal Coeur Vaiss. 2006 Sep;99(9):798-803. French. PMID 17067098
- [Background] Fourny M, Lucas AS, Belle L, Debaty G, Casez P, Bouvaist H, Francois P, Vanzetto G, Labarere J. Inappropriate dispatcher decision for emergency medical service users with acute myocardial infarction. Am J Emerg Med. 2011 Jan;29(1):37-42. doi: 10.1016/j.ajem.2009.07.008. Epub 2010 Mar 9. PMID 20825772
- [Result] Zannad F, Briancon S, Juilliere Y, Mertes PM, Villemot JP, Alla F, Virion JM. Incidence, clinical and etiologic features, and outcomes of advanced chronic heart failure: the EPICAL Study. Epidemiologie de l'Insuffisance Cardiaque Avancee en Lorraine. J Am Coll Cardiol. 1999 Mar;33(3):734-42. doi: 10.1016/s0735-1097(98)00634-2. PMID 10080475
- [Result] Delahaye F, Roth O, Aupetit JF, de Gevigney G. [Epidemiology and prognosis of cardiac insufficiency]. Arch Mal Coeur Vaiss. 2001 Dec;94(12):1393-403. French. PMID 11828925
- [Result] Schaufelberger M, Swedberg K, Koster M, Rosen M, Rosengren A. Decreasing one-year mortality and hospitalization rates for heart failure in Sweden; Data from the Swedish Hospital Discharge Registry 1988 to 2000. Eur Heart J. 2004 Feb;25(4):300-7. doi: 10.1016/j.ehj.2003.12.012. PMID 14984918
- [Result] Logeart D, Isnard R, Resche-Rigon M, Seronde MF, de Groote P, Jondeau G, Galinier M, Mulak G, Donal E, Delahaye F, Juilliere Y, Damy T, Jourdain P, Bauer F, Eicher JC, Neuder Y, Trochu JN; Heart Failure of the French Society of Cardiology. Current aspects of the spectrum of acute heart failure syndromes in a real-life setting: the OFICA study. Eur J Heart Fail. 2013 Apr;15(4):465-76. doi: 10.1093/eurjhf/hfs189. Epub 2012 Nov 27. PMID 23186936
- [Result] Logeart D. [The OFICA study of acute heart failure]. Soins. 2013 Apr;(774):35. No abstract available. French. PMID 23697057
- [Result] Nguyen HB, Rivers EP, Havstad S, Knoblich B, Ressler JA, Muzzin AM, Tomlanovich MC. Critical care in the emergency department: A physiologic assessment and outcome evaluation. Acad Emerg Med. 2000 Dec;7(12):1354-61. doi: 10.1111/j.1553-2712.2000.tb00492.x. PMID 11099425
- [Result] Sebat F, Johnson D, Musthafa AA, Watnik M, Moore S, Henry K, Saari M. A multidisciplinary community hospital program for early and rapid resuscitation of shock in nontrauma patients. Chest. 2005 May;127(5):1729-43. doi: 10.1378/chest.127.5.1729. PMID 15888853
- [Result] Masip J, Roque M, Sanchez B, Fernandez R, Subirana M, Exposito JA. Noninvasive ventilation in acute cardiogenic pulmonary edema: systematic review and meta-analysis. JAMA. 2005 Dec 28;294(24):3124-30. doi: 10.1001/jama.294.24.3124. PMID 16380593
- [Result] Peter JV, Moran JL, Phillips-Hughes J, Graham P, Bersten AD. Effect of non-invasive positive pressure ventilation (NIPPV) on mortality in patients with acute cardiogenic pulmonary oedema: a meta-analysis. Lancet. 2006 Apr 8;367(9517):1155-63. doi: 10.1016/S0140-6736(06)68506-1. PMID 16616558